CLINICAL TRIAL: NCT03920618
Title: Study on Three Types of Nucleotide/Nucleoside Analogues Treatment in Patients With Hepatitis b Virus Related Acute-on-chronic Liver Failure
Brief Title: Three Types of Nucleotide/Nucleoside Analogues Treatment in HBV Related ACLF
Acronym: HBV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL6
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B; Acute-On-Chronic Liver Failure
Keywords: hepatitis b virus; acute-on-chronic liver failure; nucleotide; nucleoside
MeSH Terms: conditions — Hepatitis B; Acute-On-Chronic Liver Failure | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ETV group (Active Comparator): 50 patients would receive treatment of oral entecavir (ETV) 0.5 mg once per day from baseline to life-long.
  Interventions: Drug: Entecavir
- TDF group (Active Comparator): 50 patients would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day from baseline to life-long.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- TAF group (Experimental): 50 patients would receive treatment of oral tenofovir alafenamide (TAF) 25 mg once per day from baseline to life-long.
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Entecavir — Patients would receive treatment of oral entecavir (ETV) 0.5 mg once per day.
  Other Names: Baraclude
  Arms: ETV group
Drug: Tenofovir Disoproxil Fumarate — Patients would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day.
  Other Names: Viread
  Arms: TDF group
Drug: Tenofovir Alafenamide — Patients would receive treatment of oral tenofovir alafenamide (TAF) 25 mg once per day.
  Other Names: Vemlidy
  Arms: TAF group

SUMMARY:
This study is to investigate the clinical efficacy of three types of nucleotide/nucleoside analogues in treatment of HBV-related acute-on-chronic liver failure.

DETAILED DESCRIPTION:
Hepatitis b virus (HBV) related acute-on-chronic liver failure (ACLF) is a serious condition with high mortality rate in China. Nucleotide/nucleoside analogues are used for anti-virus treatment in these patients. Entecavir, Tenofovir Disoproxil Fumarate and Tenofovir Alafenamide are first line drug in China. But there still lacks of data of Tenofovir Alafenamide in treatment of HBV related ACLF. This study is to investigate the clinical efficacy of three types of nucleotide/nucleoside analogues in treatment of HBV related ACLF.

ELIGIBILITY:
Inclusion Criteria:

1. Positive hepatitis b surface antigen or hepatitis b virus DNA > 0.5 year;
2. Age from 12 to 65 years old;
3. Serum total bilirubin level > 10 times upper limit of normal;
4. Prothrombin time activity < 40% or prothrombin time international ratio > 1.5；
5. Do not receive nucleotide/nucleoside analogues treatment in the past half year.

Exclusion Criteria:

1. Other active liver diseases;
2. Hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases;
6. Other important organ dysfunctions;
7. Using glucocorticoid;
8. Patients can not follow-up;
9. Investigator considering inappropriate.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate in the follow-up | 144 week
  Whether patients will survive after treatment is observed in the follow-up.

SECONDARY OUTCOMES:
Model for end-stage liver disease (MELD) score is recorded after treatment | 0 week, 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  The calculation of model for end-stage liver disease (MELD) score is: R=0.378ln[serum total bilirubin (mg/dl)]+1.12ln(prothrombin time international normalized ratio)+0.95ln[serum creatinin(mg/dl)]+0.64. The higher the MELD score, the higher the mortality rate. MELD score is recorded after treatment.
Ratio of patients with undetectable hepatitis b virus DNA after treatment | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b virus DNA would be tested to know the ratio of patients with undetectable hepatitis b virus DNA at 7 time points after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang Y, Xu W, Deng Z, Wang L, Zheng X, Zhu X, Li X, Li J, Shu X, Lai J, Peng L, Xie C. Long-term efficacy and safety of tenofovir alafenamide, tenofovir disoproxil fumarate, and entecavir in treating hepatitis B virus-related acute-on-chronic liver failure: A 144-week data analysis. Liver Res. 2024 Oct 24;8(4):295-303. doi: 10.1016/j.livres.2024.10.001. eCollection 2024 Dec. PMID 39958923